CLINICAL TRIAL: NCT02197520
Title: The Effect of Treatment With Basal Insulin Peglispro or Insulin Glargine on Insulin Sensitivity and the Effect of Prandial Insulin Lispro in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study To Compare the Effects of Insulin Peglispro and Glargine on Insulin Sensitivity and Meal Time Insulin Requirements in Type 2 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15407; I2R-MC-BIDV (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — basal insulin peglispro; LY2605541; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Peglispro (with Insulin Lispro) (Experimental): Insulin peglispro, a once daily subcutaneous(SC) injection at bedtime for 5 weeks
  Interventions: Drug: Insulin Peglispro; Drug: Insulin Lispro
- Insulin Glargine (with Insulin Lispro) (Active Comparator): Insulin glargine, a once daily subcutaneous(SC) injection at bedtime for 5 weeks
  Interventions: Drug: Insulin Glargine; Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Peglispro — Administered subcutaneously (SC), (U-100 formulation)
  Other Names: LY2605541
  Arms: Insulin Peglispro (with Insulin Lispro)
Drug: Insulin Glargine — Administered subcutaneously (SC), (U-100 formulation)
  Arms: Insulin Glargine (with Insulin Lispro)
Drug: Insulin Lispro — Administered subcutaneously (SC), (U-100 formulation)

SUMMARY:
This study will look into insulin sensitivity (how the body responds to insulin) and effects of meals on type 2 diabetics comparing insulin peglispro to insulin glargine. The study has two treatment periods, each of which will last about four weeks. One drug (insulin peglispro or insulin glargine) will be administered in each period. Participants will receive both drugs during the study. Participants may remain on stable dose metformin, as prescribed by their personal physician.

ELIGIBILITY:
Inclusion Criteria:

* Stable glycated hemoglobin (HbA1c) less than (<) 10.0 percent (%)
* Stable dose of either 0.2 to 1.5 units per kilogram per day (U/kg/day) basal insulin or a total daily insulin dose l<2.0 units per kilogram (U/kg)
* C-peptide <0.3 nanomole per liter (nmol/L)
* Stable body during the last 2 months

Exclusion Criteria:

* Corrected QT interval (QTc) prolongation greater than (>) 500 milliseconds (ms) or have any other abnormality in the 12 lead
* Abnormal blood pressure
* A history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (apart from Type 1 Diabetes Mellitus (T1DM)), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Currently treated with oral antidiabetic drugs (OADs) (excluding metformin and dipeptidyl peptidase-4 (DPP4) inhibitors), or glucagon-like peptide-1 (GLP-1) agonists or intend to use over-the counter or prescription medication, herbal medications, or nutritional supplements that affect PG or insulin sensitivity, impact on hypoglycemic awareness or promote weight loss within 4 weeks prior to randomization
* Fasting triglycerides (TGs) >400 milligrams per deciliter (mg/dL) (4.52 millimoles per liter (mmol/L))
* Have used systemic or inhaled corticosteroids/glucocorticoid therapy (excluding topical, intra-articular, and intraocular preparations) within 4 weeks prior to randomization
* Currently receive insulin by pump or insulin degludec
* Poorly controlled diabetes or known to have poor awareness of hypoglycemia
* History of gastroparesis or gastrointestinal malabsorption
* Require treatment with any drug other than insulin to treat diabetes
* Previous history of proliferative retinopathy
* Excessive consumers of xanthines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institute for Clinical Research Inc, Chula Vista, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence AB: A: Insulin peglispro, administered SC for 33 days B. Insulin glargine, administered SC for 33 days
- Sequence BA: B. Insulin glargine, administered SC for 33 days A: Insulin peglispro, administered SC for 33 days
Period: Period 1
Arm/Group | Sequence AB | Sequence BA
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | Sequence AB | Sequence BA
Started | 11 | 12
Completed | 10 | 10
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- All Participants: All participants who received Insulin peglispro, administered SC for 33 days then Insulin glargine, administered SC for 33 days or Insulin glargine, administered SC for 33 days then Insulin peglispro, administered SC for 33 days
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics (PD): Average Glucose Infusion Rate From Euglycemic 2-step Hyperinsulinemic Clamp (M-value)
Description: During the euglycemic 2-step hyperinsulinemic clamp, both low and high insulin was infused sequentially during the same procedure. The 2-step clamp procedure allowed insulin sensitivity to be measured in participants and uses a lower dose of insulin of which the effect is largely on the liver and a high dose of insulin at which the effect has reached 100% on liver and effects are largely on glucose uptake in peripheral tissues. Measurements for average glucose infusion rate are collected for both steps (low and high) of the clamp procedure.
Time Frame: Day 33, last 30 minutes (final step) of euglycemic 2-step hyperinsulinemic clamp
Population: All participants who received at least 1 dose of study drug and had evaluable PD parameters.
Measure: Mean (Standard Deviation); unit: milligram*hour per deciliter
Groups:
- Insulin Peglispro: Insulin peglispro, a once daily SC
- Insulin Glargine: Insulin glargine, a once daily SC
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 21 | 22
milligram*hour per deciliter
  High Dose Insulin | 59.09 (10.48) | 55.52 (16.50)
  Low Dose Insulin | 17.22 (6.24) | 19.67 (7.61)

2. Secondary Outcome: Pharmacodynamics (PD): Plasma Glucose Area Under the Concentration Curve Zero Through 5 Hours (AUC 0-5h), Above Pre Meal Baseline for Insulin Lispro
Time Frame: Days 30 through 32:Pre-dose, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes post-breakfast
Population: All participants who received at least 1 dose of study drug and had evaluable PD parameters.
Measure: Mean (Standard Deviation); unit: milligram*hour per deciliter
Groups:
- Insulin Peglispro: Insulin peglispro, once daily SC
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 23 | 22
milligram*hour per deciliter
  10% Insulin Lispro Dose: number analyzed (Participants) | 21 | 19
  10% Insulin Lispro Dose | 437.78 (147.47) | 398.26 (159.89)
  20% Insulin Lispro Dose: number analyzed (Participants) | 21 | 18
  20% Insulin Lispro Dose | 334.23 (165.96) | 343.54 (182.13)
  30% Insulin Lispro Dose: number analyzed (Participants) | 21 | 19
  30% Insulin Lispro Dose | 244.68 (136.01) | 239.83 (175.54)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve Concentration Curve Zero Through 5 Hours (AUC 0-5h) for Prandial Insulin Lispro
Time Frame: Days 30 through 32:Pre-dose, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes post-breakfast
Population: All participants who received at least 1 dose of study drug and had evaluable PK parameters.
Measure: Mean (Standard Deviation); unit: picomol*hour per liter
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 21 | 21
picomol*hour per liter | 839 (47) | 835 (64)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve Zero Through 5 Hours (AUC 0-5h) for Acetaminophen
Time Frame: Day 29:Pre-dose, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes post-breakfast
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 23 | 22
nanograms*hour per milliliter | 33700 (28) | 35700 (31)

5. Secondary Outcome: Appetite and Satiety Ratings, as Measured Using Visual Analog Scale (VAS) on Day 29
Description: VAS was scored from 0 - 100 millimeters (mm) as a perception of appetite and satiety (Flint et al. 2000), 0 being not hungry at all or nothing at all and 100 being extremely hungry and extremely large amount.
  The questions are abbreviated in table from: How hungry do you feel right now? to Hunger and How much food do you think you could eat right now? to Food amount. Scores were averaged and will be presented and calculated by a sum of the scores dividing by the total by the number of scores reported for timepoints.
Time Frame: Day 29:Upon waking, pre-breakfast, 1 hour (hr), 2 hr, 3 hr, 4 hr and 5 hr post breakfast
Population: All participants who received at least 1 dose of study drug and had a VAS score.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 21 | 21
millimeters
  Hunger: Waking | 25.7 (23.2) | 38.6 (31.3)
  Food amount: Waking | 30.2 (23.9) | 34.4 (25.6)
  Hunger: Pre-breakfast | 41.5 (30.1) | 51.4 (32.8)
  Food amount: Pre-breakfast | 43.9 (27.7) | 51.5 (30.2)
  Hunger: 1 hour Post-breakfast | 7.8 (12.8) | 6.2 (16.4)
  Food amount: 1 hour Post-breakfast | 8.7 (12.2) | 6.0 (11.6)
  Hunger: 2 hour Post-breakfast | 19.7 (23.5) | 14.9 (19.4)
  Food amount: 2 hour Post-breakfast | 20.7 (24.2) | 16.3 (17.4)
  Hunger:3 hour Post-breakfast | 34.8 (26.5) | 29.2 (20.8)
  Food amount: 3 hour Post-breakfast | 35.6 (27.3) | 31.1 (20.6)
  Hunger: 4 hour Post-breakfast | 46.6 (27.8) | 48.0 (28.3)
  Food amount: 4 hour Post-breakfast | 48.2 (27.5) | 48.5 (28.2)
  Hunger: 5 hour Post-breakfast | 56.8 (28.6) | 55.5 (34.1)
  Food amount: 5 hour Post-breakfast | 57.5 (27.2) | 53.4 (34.4)

6. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) for Insulin Lispro During Clamp
Time Frame: Day 33 during euglycemic 2-step hyperinsulinemic clamp
Population: No participant analyzed because Outcome Measure was incorrectly registered.
Groups:
- Insulin Glargine: Insulin peglispro, a once daily SC
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Insulin Peglispro | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 14/24 | 10/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=24) | Insulin Glargine (N=23)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Catheter site haemorrhage (General disorders) | 2 (2) | 1 (1)
Catheter site related reaction (General disorders) | 3 (3) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 2 (3)
Vessel puncture site bruise (General disorders) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (6)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days